CLINICAL TRIAL: NCT04152694
Title: Ceftaroline Pharmacokinetics in Critically Ill Patients Receiving Continuous Renal Replacement Therapy
Brief Title: Ceftaroline Pharmacokinetics in Continuous Renal Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mojdeh Heavner, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00077498
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Infection During Renal Replacement Therapy; Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ceftaroline in CRRT (Other): Ceftaroline levels measured in patients receiving continuous renal replacement therapy
  Interventions: Other: Ceftaroline levels in CRRT

INTERVENTIONS:
Other: Ceftaroline levels in CRRT — Levels of ceftaroline measured in patients receiving CRRT

SUMMARY:
Dosing of ceftaroline in patients with chronic kidney disease is defined, but there is no data on pharmacokinetics and pharmacodynamics of the drug in patients receiving continuous renal replacement therapy (CRRT). The purpose of this study is to determine pharmacokinetics and pharmacodynamics of ceftaroline in a critically ill patient population receiving CRRT, in order to define a dosing recommendation in this population.

DETAILED DESCRIPTION:
Ceftaroline fosamil is a time-dependent, hydrophilic, bactericidal fifth generation cephalosporin that was FDA approved in 2010 for community acquired pneumonia and skin and skin structure infections. Ceftaroline is FDA approved for both Gram-positive and Gram-negative organisms. Gram-positive organisms covered are Staphylococcus aureus (methicillin resistant and methicillin sensitive strains), Streptococcus agalactiae, Streptococcus pneumonia, and Streptococcus pyogenes. Gram-negative coverage includes Escherichia coli, Haemophilus influenza, Klebsiella pneumonia, and Klebsiella oxytoca. In order for ceftaroline to exhibit effective bacterial killing, it requires that a certain percentage of the dosing interval is spent above the MIC.

Dosing of ceftaroline in patients with chronic kidney disease is defined, but there is no data on pharmacokinetics and pharmacodynamics of the drug in patients receiving continuous renal replacement therapy (CRRT). The purpose of this study is to determine pharmacokinetics and pharmacodynamics of ceftaroline in a critically ill patient population receiving CRRT, in order to define a dosing recommendation in this population. CRRT modes that patients may be receiving in this trial include: continuous veno-venous hemofiltration (CVVH), continuous veno-venous hemodialysis (CVVHD), and continuous veno-venous hemodiafiltration (CVVHDF).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an intensive care unit
* Receiving CRRT (CVVH, CVVHDF, CVVHD)
* Receiving ceftaroline

Exclusion Criteria:

* Pregnant patients
* Burn patients
* Patients with toxic epidermal necrolysis or Stevens-Johnson syndrome
* Patients prescribed extended infusion ceftaroline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Ceftaroline pharmacokinetics in critically ill patients receiving continuous renal replacement therapy - Half-life | 1 year
  Ceftaroline elimination half-life
Ceftaroline pharmacokinetics in critically ill patients receiving continuous renal replacement therapy - Clearance | 1 year
  Ceftaroline clearance
Ceftaroline pharmacokinetics in critically ill patients receiving continuous renal replacement therapy - Volume of distribution | 1 year
  Ceftaroline volume of distribution
Ceftaroline pharmacokinetics in critically ill patients receiving continuous renal replacement therapy - Sieving coefficient | 1 year
  Continuous renal replacement therapy modality sieving coefficient for ceftaroline

SECONDARY OUTCOMES:
Ceftaroline pharmacodynamics in patients receiving continuous renal replacement therapy | 1 year
  Percentage of time ceftaroline levels are above the minimum inhibitory concentration for the most likely pathogen(s)

CONTACTS AND LOCATIONS:
Overall Officials: Mojdeh Heavner, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States